CLINICAL TRIAL: NCT03578783
Title: A Pilot Multicenter, Randomized, Double-Blind Study Comparing The Proportion Of Responders to PSD502 and to Placebo Using the PEBEQ In Subjects With Premature Ejaculation
Brief Title: PSD502 in Subjects With Premature Ejaculation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Plethora Solutions Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSD502-PE-008
Record Dates: First submitted 2018-06-14; First posted 2018-07-06 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PSD502 (Experimental): PSD502 spray contains a eutectic-like mixture of lidocaine and prilocaine, and a propellant (norflurane) which also serves as a solvent. Each spray contains 7.5 mg lidocaine and 2.5 mg prilocaine. A single dose consists of 3 sprays applied to the glans penis.
  Interventions: Drug: PSD502
- Placebo (Placebo Comparator): The placebo is a metered dose spray, identical in appearance to the active treatment and contains the same propellant (norflurane) but has no lidocaine or prilocaine (instead it contains PEG600 and Povidone).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — For each sexual encounter during the 4-week treatment period the study spray will be applied 5 minutes before intercourse and any excess will be wiped off prior to penetration.
  Study subjects should leave at least 24 hours between each dosing.
  Arms: Placebo
Drug: PSD502 — For each sexual encounter during the 4-week treatment period the study spray will be applied 5 minutes before intercourse and any excess will be wiped off prior to penetration.
  Study subjects should leave at least 24 hours between each dosing.
  Arms: PSD502

SUMMARY:
This study is being done to test the effect of PSD502 (the study medication) compared to placebo in subjects with premature ejaculation. PSD502 is a topical (applied to skin) anesthetic spray containing a mixture of two drugs called lidocaine and prilocaine that will be applied to the penis. Half of the subjects will receive PSD502 and half will receive placebo.

DETAILED DESCRIPTION:
The study will assess whether the bothersome symptoms of premature ejaculation (PE) are helped when treated with PSD502 by answering questionnaires such as the 'Premature Ejaculation Bothersome Evaluation Questionnaire' (PEBEQ) and 'Index of Premature Ejaculation© (IPE) and some additional questions about premature ejaculation.

The study will also measure the effect of PSD502 on the Intravaginal Ejaculatory Latency Time (IELT). This is the time between when the penis enters the vagina and when the subject starts to ejaculate in the vagina.

Subjects are stratified based on whether they are circumcised or uncircumcised and within each stratified group subjects are randomized to PSD502 (lidocaine prilocaine spray) or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Male and aged 18 years and over.
* Diagnosed with PE according to the ISSM definition, that is, he ejaculates always or nearly always prior to or within about one minute of vaginal penetration; and is unable to delay ejaculation on all or nearly all vaginal penetrations; and experiences negative personal consequences, such as distress, bother, frustration and/or the avoidance of sexual intimacy.
* Subject has lifelong PE from the first sexual experience.
* Subject must be in a stable heterosexual and monogamous relationship of at least 3 months' duration with this partner.
* Subject has at least documented 3 sexual encounters, each separated by an interval of at least 24 hours, in the baseline period.
* IELT ≤1 minute in all sexual encounters in the baseline period.
* The subject's partner must provide written informed consent, be aged 18 years or over and willing to comply with the study procedures.
* Subject indicates a level of Bother on Item 3 of the PEBEQ of either "moderately", "quite a bit" or "extremely" on all encounters during the baseline period.
* Subject registers a level of "bother" at a score of 4 or greater on an 11-point NRS scale at Screening to ensure that subjects not bothered by the quickness of their ejaculation are not entered into the baseline period.

Exclusion Criteria:

* Subject, or his sexual partner, has received an investigational (unapproved) drug within 30 days of Screening.
* Subject has erectile dysfunction, defined as an IIEF-5 score of 21, unless the low score is entirely related to PE symptoms in the opinion of the Investigator.
* The subject, or his sexual partner, has a physical or psychological condition that would prevent them from undertaking the study procedures, including, but not limited to, the following:

  1. Urological disease (e.g., prostatitis, urinary tract infection) or genitourinary surgery within 8 weeks of Screening.
  2. Ongoing significant psychiatric disorder (e.g., bipolar disease, depression / anxiety disorder or schizophrenia) not controlled by medication.
* Subject has safety testing abnormalities at the Screening Visit, in particular liver function tests or anemia, that are indicative of a medical condition that would preclude further participation in the opinion of the Investigator.
* Subjects taking tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs) or selective serotonin reuptake inhibitors (SSRIs), for indications other than PE, where the dose has been changed within 4 weeks of Screening or it is planned that the dose will change during the treatment period.
* Subject has received any treatment for PE e.g., anti-depressant therapy, local anesthetic spray, eutectic mixture of local anesthetics (EMLA®) cream, intra-cavernosal injection, tramadol or psychotherapy within 4 weeks of Screening
* Subject, or his sexual partner, has a current history of alcohol or drug abuse, in the opinion of the Investigator.
* The subject, or his sexual partner, is unlikely to understand or be able to comply with study procedures, for whatever reasons.
* Subject, or his sexual partner, has known drug sensitivity to amide-type local anesthetics.
* Subjects with pregnant partners.
* Subject with sexual partners of child-bearing potential and not using appropriate contraception (hormonal contraception or intra-uterine device [IUD]).
* Subject, or his sexual partner, has a history of glucose-6-phosphate dehydrogenase (G 6 PD) deficiency or currently using medications that would increase susceptibility to methemoglobinemia (e.g., anti-malarial agents) or has congenital or acquired methemoglobinemia, or is at risk of industrial exposure to agents causing methemoglobinemia.
* Subject, or his sexual partner, uses Class I (e.g., mexiletine, tocainide) or III (e.g., amiodarone, sotalol) anti-arrhythmic drugs, or cimetidine, beta blockers or local anesthetics.
* Subject has received PSD502 in a clinical study or has received Fortacin within 1 year of Screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change between Baseline and 4 weeks : Success on the Premature Ejaculation Bothersome Evaluation Questionnaire PEBEQ Item 3 (event-specific bother) | Baseline and 4 week treatment period
  Success is defined as having a 1-point or greater improvement between the mean response over the treatment period and the mean response during the baseline period

SECONDARY OUTCOMES:
Patient Global Impression of Change | 4 weeks post treatment
  Patient-reported global impression of change in the quickness of their ejaculation. Subjects will be asked to provide a response to the question 'Compared to when you started the study, how would you describe any change in how quickly you ejaculate now?' on a 7-point scale of: 'A great deal better', 'Moderately better', 'A little better', 'About the same', 'A little worse', 'Moderately worse' and 'A great deal worse'. Subjects will also be asked to provide a 'Yes' or 'No' response to the question 'Was this a meaningful or important change for you?'
Patient Global Impression of Severity | Baseline and 4 week treatment period
  Change from baseline in patient-reported impression of severity of the quickness of their ejaculation.Subjects will be asked to answer the question 'Overall, how severe is the quickness of your ejaculation?' using a 5-point scale of 'Not Severe', 'Mildly Severe', 'Moderately Severe', 'Very Severe' and 'Extremely Severe'.
Patient Global Impression of Change-Bother | 4 weeks post treatment
  Patient-reported global impression of change in the bother resulting from the quickness of their ejaculation. Subjects will be asked to provide a response to the following question 'Compared to when you started the study, how would you describe any change in how much you are bothered by the quickness of your ejaculation now?' on a 7-point scale of: 'Bothered a great deal less', 'Bothered moderately less', 'Bothered a little less', 'Bothered about the same', 'Bothered a little worse', 'Bothered moderately worse' and 'Bothered a great deal worse'. Subjects will also be asked to provide a 'Yes' or 'No' response to the question 'Was this a meaningful or important change for you?'.
Intravaginal ejaculatory latency time | Baseline and 4 week treatment period
  Change from baseline in intravaginal ejaculatory latency time
Independent Ejaculation Quickness Item | Baseline and 4 week treatment period
  Change from baseline in patient-reported impression of how quickly they ejaculated during each attempt of sexual intercourse
Index of Premature Ejaculation Control Domain Score | 4 weeks post treatment
  Change from baseline in the Index of Premature Ejaculation Control Domain Score. The domain is based on 4 items (score range 4-20). Low scores represent a worse value.
Index of Premature Ejaculation Distress Domain Score | 4 weeks post treatment
  Change from baseline in the Index of Premature Ejaculation Distress Domain Score. The domain is based on two items (score range 2-10). Low scores represent a worse value.
Index of Premature Ejaculation Satisfaction Domain Score | 4 weeks post treatment
  Change from baseline in the Index of Premature Ejaculation Satisfaction Domain Score. The domain is based on 4 items (score range 4-20). Low scores represent a worse value.
Independent Numeric Response Scale Bother Item | Baseline and 4 week treatment period
  Change from baseline in patient-reported assessment of bother during each attempt of sexual intercourse
Psychometric properties of the Premature Ejaculation Bothersome Evaluation Questionnaire Item 3 (event-specific bother) | 4 weeks post treatment
  Patient-reported impression of how bothered they were by how quickly they ejaculated during each attempt of sexual intercourse. Subjects will be asked to provide a response to the question 'How bothered were you by how quickly you ejaculated during the sexual intercourse you just engaged in?' on a 5-point scale of 'Not at All', 'A Little Bit', 'Moderately', 'Quite a Bit' and 'Extremely'

CONTACTS AND LOCATIONS:
Overall Officials: Jed Kaminetsky, MD, BA, Principal Investigator — Manhattan Medical Research, 215 Lexington Avenue, 21st Floor, New York, NY 10016
Locations (21):
- United States (21):
  - Achieve Clinical Research, Birmingham, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Skyline Urology, Sherman Oaks, California
  - Imagine Research of Palm Beach County, Boynton Beach, Florida
  - SunCoast Research, Miami, Florida
  - Suncoast Research Associates, Miami Lakes, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Primary Care Research, Atlanta, Georgia
  - Georgia Clinical Research, Llc, Lawrenceville, Georgia
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Mens Health Boston, Chestnut Hill, Massachusetts
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Midlantic Urology, Bala-Cynwyd, Pennsylvania
  - Advanced Clinical Research - Jordan Ridge Family Medicine, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No